CLINICAL TRIAL: NCT03365388
Title: A Validation Study of Sodium Hyaluronate in Patients With Periarthritis of Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, pengzhang, Doctor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSG-trail201703
Record Dates: First submitted 2017-12-02; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Periarthritis
MeSH Terms: conditions — Periarthritis | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: The patient was diagnosed with periarthritis of shoulder
Who Masked: Outcomes Assessor
Masking Description: The evaluation of the subjects will be conducted by the blind researchers. The IMP administration of the subjects will be conducted by non blind researchers or legal staff authorized by the principal investigator (PI)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Hyaluronate group (Experimental): Treatment of periarthritis of shoulder with Sodium Hyaluronate
  Interventions: Drug: Sodium Hyaluronate
- Aerzhi group (Active Comparator): Treatment of periarthritis of shoulder with Aerzhi
  Interventions: Drug: Aerzhi

INTERVENTIONS:
Drug: Sodium Hyaluronate — Hyaluronic acid is a component of synovial fluid. N- is glucuronic acid and N-acetylglucosamine repeating disaccharide unit form
  Arms: Sodium Hyaluronate group
Drug: Aerzhi — Sodium Hyaluronate Injection can cover and protect joint tissue, improve lubrication function, and penetrate degenerative cartilage
  Other Names: Sodium Hyaluronate Injection
  Arms: Aerzhi group

SUMMARY:
Alge as a positive control drug, in patients with periarthritis of shoulder, in a double-blind, controlled manner to study the safety and treatment of Sodium Hyaluronate

DETAILED DESCRIPTION:
Aerzhi as a positive control drug, in patients with periarthritis of shoulder, in a double-blind, controlled manner to study the safety and treatment of Sodium Hyaluronate. Once a week, continuous treatment for 5 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Based on clinical symptoms and range of motion (ROM) limitation: abduction is not more than 135 degrees, external rotation is not more than 20 degrees or the maximum internal rotation arrives at the first lumbar spinous process (the tip of the patient can touch) to diagnose the patients with periarthritis of shoulder
2. Signs and symptoms were repeated for 12 weeks or more at the time of signing informed consent (12 weeks or more)
3. At zeroth weeks, according to the pain assessment scale (NRS, range: 0-10), the subjects' self rating pain score was no less than 5 points
4. Fully informed consent signed voluntarily informed consent

Exclusion Criteria:

1. Lead to other diseases of shoulder disorders, such as acute rotator cuff tear, calcific tendinitis. If the diagnosis is necessary, the MRI scan is performed
2. Patients who are not suitable for medical treatment (e.g. patients with surgical indications)
3. Patients who received opioids before the first study of the drug
4. Patients who received the following or more treatment within 2 weeks before the first use of the drug(Bilateral or unilateral shoulder joint movement therapy/Treatment of periarthritis of shoulder with proprietary Chinese Medicine)
5. Patients who received the following or more treatment within 4 weeks before the first use of the drug(Corticosteroids were injected locally or bilaterally on either side of the shoulder or on the other side of the shoulder (bilateral or unilateral shoulder joint);Oral corticosteroids, suppositories or intravenous preparations for the treatment of glucocorticoids)
6. Treatment of shoulder joint (bilateral or unilateral) with hyaluronic acid injection within 24 weeks before the first study of the drug
7. It is diagnosed as rheumatic disease
8. Patients unable to assess their clinical manifestations
9. Skin disease or skin infection around the injection site can cause the risk of injection infection
10. Severe heart disease, renal failure, hematologic diseases, or diabetes mellitus
11. There is a history of hypersensitivity to any component in the research drug (IMP)

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Pain Rating Scale（NRS） | Fifth weeks after medication
  At fifth weeks, subjects reported changes in NRS pain scores compared to baseline

SECONDARY OUTCOMES:
The number of adverse events | Fifth weeks after medication
  The number of adverse events：Abnormal laboratory examination results，symptoms or diseases

CONTACTS AND LOCATIONS:
Overall Officials: Peixun Zhang, Doctor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yamamoto M. Sugawara S. Tsukamoto Y. Motegi M. Iwata H. Ryu J. et al. Clinical Evaluation of high molecule weight hyaluronate (NRD101) on osteoarthritis of the knee: a phase III comparative clinical study with ARTZⓇ as a clinical drug. Jpn Pharmacol Ther 1994;22:319-47.
- [Background] Kurokawa T, Oda H, Mikami Y, Katsumoto H, Clinical Evaluation of high Molecule Weight Sodium Hyaluronate (NRD101) on osteoarthritis of the knee: phase III long-term clinical study. Jpn Pharmacol Ther 1994;22:267-88.
- [Background] Yamamoto R, Tabata S, Mikasa M, Takagishi K, Clinical evaluation of high molecule sodium hyaluronate (NRD101) on periarthritis scapulohumeralis. Jpn Pharmacol Ther 1993;21:267-80.
- [Background] Yamamoto R, Tabata S, Mikasa M, Takagishi K, Nakajima M, Dose-range finding study of high molecule weight sodium hyaluronate (NRD101) on periarthritis scapulohumeralis: a multi-center, late phase II clinical study. Jpn Pharmacol Ther 1994;22:351-74.
- [Background] Yamamoto R, Tabata S, Mikasa M, Takagishi K, Nakajima M, Phase 3 comperative clinical study of high molecular weight sodium hyaluronate (NRD101) with ARTZⓇ on periarthritis scapulohumeralis. Jpn Pharmacol Ther 1994;22:289-317.
- [Background] Tanaka S, Sohen S, Yamamoto M, Komatsubara Y, Sugawara S, Matsubara T, Additional analysis for a multi-center phase II clinical study of high molecule hyaluronic acid (NRD101) on rheumatoid arthritis. Clinical rheumatology and related research 2000:12: 157-78.
- [Background] Tanaka S, Sohen S, Yamamoto M, Komatsubara Y, Sugawara S, Matsubara T, et al. Additional analysis for a multi-center phase III comparative clinical study of high molecular hyaluronic acid (NRD101) on rheumatoid arthritis. Clinical rheumatology and related research 2000;12: 179-204
- [Background] Tanaka S, Sohen S, Yamamoto M, Komatsubara Y, Sugawara S, Matsubara T, Additional analysis for a multi-center, long-term clinical study of high molecule weight hyaluronic acid (NRD101) on rheumatoid arthritis. Clinical rheumatology and related research 2000;12:213-40.
- [Background] Zhang W, Nuki G, Moskowitz RW, Abramson S, Altman RD, Arden NK, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis: part III: Changes in evidence following systematic cumulative update of research published through January 2009. Osteoarthritis Cartilage. 2010 Apr;18(4):476-99. doi: 10.1016/j.joca.2010.01.013. Epub 2010 Feb 11. PMID 20170770